CLINICAL TRIAL: NCT06276764
Title: The LINFU® U.S. Registry for the Detection of Dysplasia and Pancreatic Ductal Adenocarcinoma (PDAC) in Patients With IPMN (Intraductal Papillary Mucinous Neoplasm of the Pancreas)
Brief Title: The LINFU® U.S. Registry in Patients With IPMN (Intraductal Papillary Mucinous Neoplasm of the Pancreas)
Status: Enrolling by invitation | Type: Observational
Sponsor: Adenocyte, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Adenocyte 103
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: IPMN, Pancreatic; Pancreas Cancer; Pancreatic Cyst
MeSH Terms: conditions — Pancreatic Intraductal Neoplasms; Pancreatic Neoplasms; Pancreatic Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Slides and cell blocks made from pancreatic fluid collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients with a documented history of IPMN: Patients with a documented history of IPMN by any imaging method will undergo the LINFU® procedure.
  Interventions: Diagnostic Test: LINFU®

INTERVENTIONS:
Diagnostic Test: LINFU® — Patients will undergo low intensity non-focused ultrasound excitation of the pancreas for a total of 15 minutes. A contrast agent will be administered IV at five minute intervals. The patient will then receive a dose of secretin and the the patient's pancreatic juice will then be collected for a total of 15 minutes.

SUMMARY:
In this study, LINFU® will be evaluated in patients who have been identified with IPMN to determine if it can be used to help identify early, pancreatic ductal adenocarcinoma and its noninvasive precursor lesions (dysplasia). The study will also help determine if LINFU® results in earlier intervention, treatment and improvement in patient outcomes.

DETAILED DESCRIPTION:
Adenocyte has developed a proprietary pancreatic cancer detection method, LINFU®, (Low Intensity Non-Focused Ultrasound excitation of the pancreas) that increases the sensitivity of pancreatic juice cytology. LINFU® excitation of circulating microbubbles increases the exfoliation of pancreatic ductal cells. The sensitivity of cytological examination of the pancreatic fluid obtained by LINFU® can also be potentially enhanced by neural network-based computer-assisted analysis.

In this study, LINFU® will be evaluated in patients who have been identified with IPMN to determine if it can be used to help identify early, pancreatic ductal adenocarcinoma and its noninvasive precursor lesions (dysplasia) which are not identified with current diagnostic tests. In addition, patients identified with PDAC or precursor lesions only with LINFU® and not detected with other diagnostic tests will be followed long term to determine the progression rate of these tumors and whether LINFU® results in earlier intervention, treatment and improvement in patient outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Both males and females will be enrolled and must be at least 18 years of age and under age of 90
2. Patients with a documented history of IPMN by any imaging method.
3. All patients must undergo contemporaneous imaging (within 90 days before or after the LINFU® procedure) with one or more of the following: EUS, CH-EUS, CEUS, MRI/MRCP, PET/CT, CT
4. Patients undergoing EUS-FNA may be enrolled but the FNA must be performed after the LINFU® procedure
5. Institutional Review Board (IRB)-approved consent must be signed by patients to participate in this study.

Exclusion Criteria:

1. Patient under the age of 18 and over the age 90
2. Contraindications to LINFU® as determined by study investigators:

   1. Patient with uncorrectable coagulopathy
   2. Patient that cannot undergo anesthesia due to cardiopulmonary contraindication as deemed by the anesthesiologist
   3. Unstable medically (cardiopulmonary, neurologic, or cardiovascular status)
3. Patients with IPMN that has been subjected to FNA or biopsy prior to the LINFU procedure
4. Patients with pancreatic cystic neoplasms other than IPMN i.e. mucinous cystic neoplasms, serous cystic neoplasms and other rare cystic lesions
5. Pregnant females will be excluded
6. Patient that is unable to provide informed consent
7. Patient with known allergy to the microbubble contrast agent or secretin

Study Design Overview:

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a documented history of IPMN by any imaging method.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2034-09-30 (Estimated); Study Completion 2034-12-01 (Estimated)

PRIMARY OUTCOMES:
The number of pancreatic ductal adenocarcinomas or their precursor lesions, dysplasia, identified only with LINFU® will be compared to standard screening methods | 5 years
  The total number of asymptomatic pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified with LINFU® by analysis of pancreatic fluid will be compared to the number of these lesions identified with current screening tests, including EUS, CH-EUS, CEUS, MRI/MRCP, PET/CT, CT

SECONDARY OUTCOMES:
The change in size of pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified only with LINFU® will be determined over a 5 year period | 5 years
  Patients with early pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified only with LINFU® and not detected with other diagnostic tests will be monitored long- term (5 years) by EUS, CH-EUS, CEUS, MRI/MRCP, PET/CT, CT to assess whether these tumors increase in size (measured in mm) and to determine how many require medical or surgical intervention.
Determine the number of patients with early pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified only with LINFU® that require medical or surgical intervention. | 5 years
  Patients with early pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified only with LINFU® and not detected with other diagnostic tests will be monitored long- term (5 years) by EUS, CH-EUS, CEUS, MRI/MRCP, PET/CT, CT to assess whether these tumors increase how many require medical or surgical intervention.

OTHER OUTCOMES:
Yearly survival rate of patients with early pancreatic ductal adenocarcinomas or their noninvasive precursor lesions identified only with LINFU® | 5 years
  Patients will be followed by EUS, CH-EUS, CEUS, MRI/MRCP, PET/CT, CT and yearly survival rates of patients with early pancreatic ductal adenocarcinomas and their noninvasive precursor lesions identified only with LINFU® and not detected with other diagnostic tests will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Haber, MD FRCP, Principal Investigator — Manhattan Endoscopy Center
Locations (1):
- Manhattan Endoscopy Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No